CLINICAL TRIAL: NCT05918614
Title: A Phase 1, Placebo-Controlled, Double-Blind Study to Examine the Safety, Tolerability, and Pharmacokinetics of 500 mg KD025 Administered Twice Daily in Healthy Male and Post-Menopausal Female Subjects
Brief Title: A Study to Determine the Effect of 500 mg Oral Dose of KD025 in Healthy Male and Post-menopausal Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kadmon, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: KD025-103; U1111-1290-9655 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06-14

CONDITIONS: Immune System Disorder (Healthy Volunteer)
MeSH Terms: conditions — Immune System Diseases | interventions — KD025

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- KD025 (Experimental): 500 mg KD025 administered orally twice daily (BID) for 28 days
  Interventions: Drug: Belumosudil mesylate
- Placebo (Placebo Comparator): Placebo administered orally BID for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Belumosudil mesylate — Pharmaceutical form: capsule; Route of administration: oral
  Other Names: KD025; SAR445761
  Arms: KD025
Drug: Placebo — Pharmaceutical form: capsule; Route of administration: oral
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and pharmacokinetics of 500 mg oral BID dose of KD025 in healthy male and post-menopausal female participants.

DETAILED DESCRIPTION:
Up to approximately 58 days including safety follow up period of 30 days after participant is treated with the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants between the ages of 18 and 55 years, inclusive.
* Female who is not of reproductive potential.
* Able to provide written informed consent prior to the performance of any study specific procedures.
* Body mass index (BMI) range of 19-30 kilogram per square meter (kg/m2), inclusive.

Exclusion Criteria:

* Past or present disease that is judged by the investigator to have the potential to interfere with the study procedures, compromise safety, or affect the PK evaluations.
* Known sensitivity to Rho-associated coiled-coil containing serine/threonine protein kinases (ROCK2) inhibitor agents or to any of the constituents of the KD025 formulation.

The above information is not intended to contain all considerations relevant to the potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2014-03-28 (Actual); Primary Completion 2014-06-07 (Actual); Study Completion 2014-06-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events and serious adverse events | Up to approximately 58 days
  Number of participants with adverse events and serious adverse events

SECONDARY OUTCOMES:
Cmax of KD025 and its metabolites [M1 (KD025m1) and M2 (KD025m2)] | Predose and multiple timepoints up to 30 hours postdose on Days 1 and 28
  Cmax maximum plasma concentration determined directly from the concentration time profile
Tmax of KD025 and its metabolites [M1 (KD025m1) and M2 (KD025m2)] | Predose and multiple timepoints up to 30 hours postdose on Days 1 and 28
  tmax, observed time to reach peak plasma concentration
Cmin of KD025 and its metabolites [M1 (KD025m1) and M2 (KD025m2)] | Predose and multiple timepoints up to 30 hours postdose on Days 1 and 28
  Cmin, Minimum or "trough" plasma concentration after its administration and just prior to the administration of a subsequent dose as determined from the concentration time cprofile
AUC0 -τ of KD025 and its metabolites [M1 (KD025m1) and M2 (KD025m2)] | Predose and multiple timepoints up to 30 hours postdose on Days 1 and 28
  AUC0 -τis area under the plasma concentration-time curve from predose (time 0) to end of dosing collection (30 hours)
AUCinf of KD025 and its metabolites [M1 (KD025m1) and M2 (KD025m2)] | Predose and multiple timepoints up to 30 hours postdose on Days 1 and 28
  AUCinf, area under the concentration-time curve from predose (time 0) extrapolated to Infinity
Accumulation ratio (R) of KD025 and its metabolites [M1 (KD025m1) and M2 (KD025m2)] | Predose and multiple timepoints up to 30 hours postdose on Days 1 and 28
  Accumulation ratio, determined as the ratio of Day 28 AUC divided by Day 1 AUC and as the ratio of Day 28 Cmax divided by Day 1 Cmax
t1/2 of KD025 and its metabolites [M1 (KD025m1) and M2 (KD025m2)] | Predose and multiple timepoints up to 30 hours postdose on Days 1 and 28
  t1/2 terminal elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational site, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org